CLINICAL TRIAL: NCT03665584
Title: A Double Blinded Sham Controlled Trial of Fractional CO2 Laser Treatment Using the DEKA SmartXide Touch Laser System (MonaLisa Touch) for the Treatment of Vulvar Lichen Sclerosus
Brief Title: MonaLisa Touch Laser for the Treatment of Vulvar Lichen Sclerosus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Vulvovaginal Disorders (Other)
Collaborators: Gynecologic Cancer Research Foundation (Other); El. En. SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00024516
Record Dates: First submitted 2018-08-06; First posted 2018-09-11 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Lichen Sclerosus
Keywords: Lichen Sclerosus; MonaLisa Touch
MeSH Terms: conditions — Lichen Sclerosus et Atrophicus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- FxCO2 Laser (Active Comparator): FxCO2 laser treatment will be performed by scanning across the entire affected anogenital region. The FxCO2 treatment will be performed at baseline and then repeated at 4 week intervals for a total of 5 treatments. The laser parameters change with each treatment: power (18, 20, 22, 24, 26W), dwell time (800, 900, 1000, 1000, 1000us) and spacing (1200, 1100, 1000, 1000, 1000um) in respective order.
  Interventions: Device: FxCO2 Laser
- Sham Laser (Sham Comparator): Sham laser treatment will be performed by scanning across the entire affected anogenital region. The sham treatment will be performed using 4W (power), 400us (dwell time), and 1500um (spacing). The laser has no effect on the vulvar tissue using these parameters.
  Interventions: Device: Sham Laser

INTERVENTIONS:
Device: FxCO2 Laser — The FxCO2 laser allows a microablative effect in soft tissue.
  Arms: FxCO2 Laser
Device: Sham Laser — The Sham laser will be used on the participants who receive the sham treatment.
  Arms: Sham Laser

SUMMARY:
Lichen sclerosus (LS) is a skin condition of the external genitals (vulva) of women. LS causes vulvar itching, pain, and burning. In addition, LS causes scarring of the vulva which may cause significant sexual dysfunction or pain. Lastly, 4-6% of women with LS will develop vulvar cancer.

The current "gold standard" treatment for lichen sclerosus is potent steroids creams. When used correctly, steroid creams help to decrease the symptoms of itching and burning and can prevent further vulvar scarring. In addition, proper treatment reverses the underlying inflammation of LS, and may lower the risk of getting cancer. While useful, steroid creams may have serious side effects that include thinning of the skin, fungal infections, and lowering the immune system.

Recently, microablative fractional CO 2 laser treatment (FxCO 2 ) (SmartXide 2 V 2 LR laser system, for MonaLisa Touch, DEKA, Florence, Italy) has been proposed for the management of LS. Specifically, two small studies demonstrated that FxCO 2 therapy appears to be a promising treatment modality to treat lichen sclerosus. These studies demonstrated that FxCO 2 treatment may stimulate tissue healing in LS. Furthermore, by reducing inflammation, the clinical symptoms of LS, such as intense itching and burning, were improved. While these studies showed good success, these studies were limited because of their small size and lack of sham (fake treatment) control.

The purpose of this study is to look at the efficacy (how well it works) and the safety of the FxCO 2 laser treatment (laser energy emitted) for LS as compared to a sham treatment (very minimal laser energy will be emitted).

DETAILED DESCRIPTION:
Lichen sclerosus (LS) is a chronic cutaneous disorder affecting approximately one in seventy women. Presenting symptoms may include intense pruritus, pain, burning, and severe dyspareunia. This disorder may affect any area of the skin, but has a notable predilection for the anogenital skin. Extra-genital involvement is infrequent, affecting only 11% of women with LS. Affected females outnumber affect males by 10:1. There is bimodal peak incidence in premenarchal girls and menopausal women with an average age of onset of 51 years of age.

The typical lesions of LS are white plaques and papules, often with areas of ecchymosis, excoriation, and ulceration. Often, there is destruction of the vulva architecture with scarring of the clitoral prepuce, resorption of the labia minora, and narrowing of the introitus. Four to six percent of women with LS will develop vulvar carcinoma. The histopathologic changes of LS are distinctive and make biopsy a very useful diagnostic tool. Characteristic pathologic finding include hyperkeratosis of the epidermis, epidermal atrophy with loss of rete ridges, homogenization of the collagen in the upper dermis, and a lichenoid (band-like) inflammatory infiltrate in the dermis. While there is no known cure for LS, the current gold standard treatment is ultra-potent corticosteroids. When properly administered, topical ultra-potent corticosteroids help to resolve the symptoms of pruritus and burning and can prevent further vulvar scarring. In addition, proper treatment reverses the underlying histopathologic changes of LS, and preliminary data shows that the risk of malignant transformation also declines.

Although treatment with topical corticosteroids is effective, topical corticosteroids may have serious local and systemic side effects, including dermal thinning, skin atrophy, superimposed infections, rebound dermatitis, and adrenal insufficiency. Due to these side effects, long- term use of corticosteroids for the treatment of vulvar lichen sclerosus may be inadvisable. Therefore, a safe and effective alternative intervention is needed for this disorder.

Recently, microablative fractional CO 2 laser (SmartXide 2 V 2 LR CO 2 laser system, for MonaLisa Touch, DEKA, Florence, Italy) has been proposed for the management of LS. This type of laser has a wavelength of 10,600 nm that allows a superficial microablative effect in soft tissues and a pulsed beam that protects the tissues from possible overheating damage. The laser beam is delivered to the tissue in a fractional manner, creating small spots (called DOTs) alternating parts of tissue treated and not treated. The size of each DOT is set by the manufacturer at 150 - 200 μm. Moreover, it has a DEKA pulse (D-pulse) mode that consists of two parts: (a) constant, high energy peak power, for rapid superficial evaporation of the atrophic epithelium with low water content and (b) lower peak power with longer emission times that allows the energy heat to penetrate deeper in the epithelium. This D-pulse mode combined with DOTs remodels the connective tissue via the production of heat shock protein 47 and produces new collagen/fibroblasts and ground matrix.

Recently, two small studies demonstrated that fractional CO 2 laser (FxCO 2 ) therapy appears to be a promising treatment modality to treat lichen sclerosus. These studies demonstrated that FxCO 2 treatment may stimulate protein synthesis, accelerate tissue reconstruction, and decrease lichenification. Furthermore, after elimination of local inflammation, the stimulus of nerve endings was reduced, so the clinical manifestations of LS, such as intense vulvar pruritus and burning were improved.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 years or older.
* Have a diagnosis of active lichen sclerosus (Dr. Goldstein will remove a pea size amount of skin (a biopsy) and will do a physical assessment of the vulva area at the beginning of the study to confirm this diagnosis).
* Are willing and able to comply with the study requirements.
* Have a negative pregnancy test prior to enrolling in this study and will use at least one form of birth control during the course of the study if you are sexually active and are of child bearing potential.
* Have at least a 3 out of 10 on a questionnaire that measures the amount of itching you are having.

Exclusion Criteria:

* Are immunocompromised (have a lowered immune system) (for example, you have been diagnosed with or have a history of lymphoma, AIDS, or Wiskott-Aldrich Syndrome), or have an uncontrolled malignant disease.
* Have a generalized infection (bacterial, viral or fungal), or obvious localized infections in the vulva area.
* Have swollen lymph nodes (lymphadenopathy).
* Have any active sexually transmitted diseases on the vulva (herpes, molluscum, condyloma).
* Have been diagnosed with other vulvar dermatologic conditions including lichen planus, psoriasis, lichen simplex chronicus, candidiasis, intraepithelial neoplasia, or carcinoma.
* Are pregnant or breastfeeding.
* If you become pregnant while on the study, you must withdraw from the study.
* Have received an investigational drug within four weeks prior to the study or who plan to use other investigational drugs during the course of this study.
* Have severe medical condition(s) that in the view of the study doctor prohibits participation in the study.
* Have a history of substance abuse or any factor, which limits your ability to cooperate with the study procedures.
* Are uncooperative or are not willing to attend regular visits.
* Have received systemic immunosuppressants (steroids), other systemic therapies or any other systemic therapies known or suspected to have an effect on vulvar lichen sclerosus within 4 weeks prior to participation in the study.
* Have been treated with topical therapy (for example, topical corticosteroids, pimecrolimus, tacrolimus) or any other topical therapies known or suspected to have an effect on vulvar lichen sclerosus or its symptoms within 4 weeks prior to participation in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-07-14 (Actual)

PRIMARY OUTCOMES:
Inflammatory Infiltration | 26 weeks
  A blinded dermatopathologist will evaluate the inflammatory infiltration on biopsy specimens obtained during screening process and after 24-week treatment period.

SECONDARY OUTCOMES:
Changes from Baseline in Clinical Scoring System for Vulvar Lichen Sclerosus | 26 weeks
  A validated scoring system will assess both the investigator's impression of the severity of the disease and the patient's impression of the severity of her disease at weeks 0, 14, and 26.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Goldstein, MD, Principal Investigator — The Centers for Vulvovaginal Disorders
Locations (1):
- The Centers for Vulvovaginal Disorders, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mitchell L, Goldstein AT, Heller D, Mautz T, Thorne C, Joyce Kong SY, Sophocles ME, Tolson H, Krapf JM. Fractionated Carbon Dioxide Laser for the Treatment of Vulvar Lichen Sclerosus: A Randomized Controlled Trial. Obstet Gynecol. 2021 Jun 1;137(6):979-987. doi: 10.1097/AOG.0000000000004409. PMID 33957648